CLINICAL TRIAL: NCT02905526
Title: A Randomised Controlled Trial of an Intervention Delivered by App Instant Messaging to Increase Use of Effective Contraception Among Young Women in Bolivia
Brief Title: An Intervention Delivered by App Instant Messaging to Increase Use of Effective Contraception Among Young Women in Bolivia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: International Planned Parenthood Federation (Other); Centro de Investigacion, Educacion y Servicios (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10999
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2017-09

CONDITIONS: Contraception
Keywords: Reproductive health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): App plus the contraceptive instant messages
  Interventions: Behavioral: Contraceptive instant messages; Other: Mobile phone app
- Control (Placebo Comparator): App only
  Interventions: Other: Mobile phone app

INTERVENTIONS:
Behavioral: Contraceptive instant messages — Contraceptive Instant messages
  Arms: Intervention
Other: Mobile phone app — Mobile phone app

SUMMARY:
This randomised controlled trial will establish the effect a contraceptive intervention delivered by mobile phone app instant messaging on use of effective contraception in Bolivia. Woman aged 16-24 will be randomised to have access to Centro de Investigacion, Educacion y Servicios's sexual and reproductive health app (control) or the app plus 0-3 instant messages a day for 4 months (intervention). Participants will complete a questionnaire at baseline and 4 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-24
* Own a personal Android mobile phone
* Live in El Alto or La Paz Bolivia
* Sexually active
* Not using the pill, implant, injection, intrauterine device or patch
* Want to avoid a pregnancy

Exclusion Criteria:

* Cannot read Spanish

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 645 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Use of effective contraception | 4 months
  The proportion reporting current use of effective contraception (pill, intrauterine device, injection, implant, patch)
Acceptability of at least one method of effective contraception | 4 months
  The proportion reporting that at least one method of effective contraception is acceptable (pill, intrauterine device, injection, implant, patch)

SECONDARY OUTCOMES:
Acceptability of individual effective contraceptive methods | 4 months
  The proportion reporting that individual methods of effective contraception are acceptable (pill, intrauterine device, injection, implant, patch)
Discontinuation of effective contraception | 4 months
  The proportion reporting use of effective contraception at any time during the 4 months (pill, intrauterine device, injection, implant, patch)
Service uptake | 4 months
  The proportion reporting attending a sexual health service during the 4 months
Unintended pregnancy | 4 months
  The proportion reporting that they became pregnant and did not want to become pregnant during the study
Induced abortion | 4 months
  The proportion reporting having an abortion during the study

OTHER OUTCOMES:
Knowledge of effective contraception | 4 months
  Score on the knowledge measure
Perceived norms in relation to using and communicating with partners about contraception | 4 months
  Responses to the perceived norms scales
Personal agency in using and communicating with partners about contraception | 4 months
  Responses to the personal agency scales
Intention to use effective contraception | 4 months
  Response to the intention scale
Intervention 'dose' received | 4 months
  If participants read all, some, most or none of the messages and if they stopped the messages

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Free, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Centro de Investigacion, Educacion y Servicios, La Paz, Bolivia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McCarthy OL, Aliaga C, Torrico Palacios ME, Lopez Gallardo J, Huaynoca S, Leurent B, Edwards P, Palmer M, Ahamed I, Free C. An Intervention Delivered by Mobile Phone Instant Messaging to Increase Acceptability and Use of Effective Contraception Among Young Women in Bolivia: Randomized Controlled Trial. J Med Internet Res. 2020 Jun 22;22(6):e14073. doi: 10.2196/14073. PMID 32568092
- [Derived] McCarthy OL, Osorio Calderon V, Makleff S, Huaynoca S, Leurent B, Edwards P, Lopez Gallardo J, Free C. An Intervention Delivered by App Instant Messaging to Increase Acceptability and Use of Effective Contraception Among Young Women in Bolivia: Protocol of a Randomized Controlled Trial. JMIR Res Protoc. 2017 Dec 18;6(12):e252. doi: 10.2196/resprot.8679. PMID 29254910